CLINICAL TRIAL: NCT02671474
Title: Valve Leaflet Motion in Sutureless Bioprosthetic Aortic Valves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, Karolinska University Hospital
Purpose: Diagnostic
Other Study IDs: Perceval thrombosis
Record Dates: First submitted 2016-01-24; First posted 2016-02-02 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Aortic Valve Stenosis; Heart Valve Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

INTERVENTIONS:
Other: 4-dimensional volume-rendered computed tomography

SUMMARY:
A single-center prospective interventional trial. Patients implanted with a sutureless bioprosthetic aortic valve at Karolinska University Hospital in Stockholm, Sweden from 2012 will be eligible. 4-dimensional volume-rendered computed tomography (CT) of the heart will be performed. The aim of the CT is to assess valve leaflet motion. Results of the CT examination, preoperative clinical characteristics, and postoperative clinical data will be registered. Data will be collected prospectively and retrospectively. Informed consent will be obtained from patients meeting the inclusion criteria before the initiation of any study-specific procedures.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a sutureless Perceval (Sorin Group) sutureless bioprosthetic aortic valve at Karolinska University Hospital in Stockholm, Sweden between 2012 and 2016
* Provide written informed consent

Exclusion Criteria:

* Contraindication for CT with intravenous contrast injection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduced aortic valve leaflet motion | At CT performed once no less than 30 days and up to 10 years after aortic valve replacement

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery and Anesthesiology, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Dalen M, Sartipy U, Cederlund K, Franco-Cereceda A, Svensson A, Themudo R, Svenarud P, Bacsovics Brolin E. Hypo-Attenuated Leaflet Thickening and Reduced Leaflet Motion in Sutureless Bioprosthetic Aortic Valves. J Am Heart Assoc. 2017 Aug 21;6(8):e005251. doi: 10.1161/JAHA.116.005251. PMID 28862959